CLINICAL TRIAL: NCT03409874
Title: Dry Needling and Spinal Manipulation or Interocclusal Appliance (Splint), NSAIDs and Joint Mobs for Temporomandibular Dysfunction
Brief Title: Dry Needling and Spinal Manipulation vs. Interocclusal Appliance (Splint), NSAIDs and Joint Mobs for Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Principal Investigator, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT16
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Dry Needling; Manipulation, Spinal; Splints; Anti-Inflammatory Agents, Non-Steroidal; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling and Spinal Manipulation (Experimental)
  Interventions: Other: Dry Needling; Other: Spinal manipulation
- Interocclusal Appliance, NSAIDs and TMJ Mobs (Active Comparator)
  Interventions: Other: Interocclusal Appliance; Drug: NSAIDs; Other: TMJ Mobs

INTERVENTIONS:
Other: Dry Needling — Dry needling to the muscle of mastication and temporomandibular joint capsule. 1-2 treatment sessions per week for up to 4 weeks
  Arms: Dry Needling and Spinal Manipulation
Other: Spinal manipulation — Spinal manipulation, targeting the upper cervical spine (C1-C2, C2-C3 or OA). 1-2 treatments per week for up to 4 weeks.
  Arms: Dry Needling and Spinal Manipulation
Other: Interocclusal Appliance — Interocclusal appliance worn every nights for 4 weeks.
  Other Names: splint
  Arms: Interocclusal Appliance, NSAIDs and TMJ Mobs
Drug: NSAIDs — diclofenac (Voltaren) 3 X 50mg per day for 4 weeks. If the patient's TMJ pain improves, the dosage may be reduced to 2 X 50mg per day.
  Other Names: diclofenac; Voltaren
  Arms: Interocclusal Appliance, NSAIDs and TMJ Mobs
Other: TMJ Mobs — Temporomandibular joint mobilization targeting the temporomandibular joint capsule. 1-2 treatments per week for up to 4 weeks.
  Arms: Interocclusal Appliance, NSAIDs and TMJ Mobs

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with temporomandibular dysfunction (TMD): Dry needling and spinal manipulation or Interocclusal Appliance (Splint), NSAIDs and Temporomandibular Joint Mobilization . Clinicians commonly use all of these techniques to treat TMD. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with stress temporomandibular dysfunction will be randomized to receive 1-2 treatment sessions per week for up to 4 weeks ( up to 8 sessions total) of either: (1) dry needling and spinal manipulation or (2) Interocclusal appliance (splint), NSAIDs, temporomandibular joint mobilization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old
2. Patient referred to physical therapy from a physician or dentist with a diagnosis of temporomandibular dysfunction that is consistent with the Revised TMD Group 1 Muscle Disorders Diagnostic Algorithm. (Dworkin et al.1992; Look et al., 2010]. According to Blanco-Hungria et al. (2015), this category represents 88.7% of patients with TMD.
3. History of symptoms related to TMD for at least 3 months
4. Intensity of pain related to TMD at least 30mm out 100 per Visual Analogue scale (La Touche et al, 2009; Gonzalez-Ingesias et al., 2013)
5. Patient presents with the following: (Gonzalez Perez et al., 2015)

   1. Strong pain in the anterior part of the lower belly of the LPM on palpation
   2. Deep-seated pain in the TMJ and/or region of the maxillary sinus (referred pain)
   3. Significant motor dysfunction (e.g. limited jaw opening, painful protrusion of the chin against resistance, mandibular lateralization to the opposite side upon opening).

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: severe hypertension, infection, ankylosing spondylitis, neoplasm, uncontrolled diabetes, peripheral neuropathy, heart disease, stroke, chronic, ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. Signs or symptoms of disc displacement, arthrosis or arthritis of the temporomandibular joint according to category II and III of the Research Diagnostic Criteria for Temporomandibular Disorders
3. History of traumatic injury such as a fracture or whiplash
4. Concomitant diagnosis of any primary headache (i.e. tension type headache or Migraine) except cervicogenic headaches
5. History of surgery related to TMD
6. Diagnosis of fibromyalgia
7. Systemic disease such as RA, lupus erythematosus or psoriatic arthritis
8. Presence of neurological disorder such as trigeminal neuralgia
9. History of PT, acupuncture or splint treatment within 3 months of the study
10. History of taking prescription NSAIDs within 3 months of the study
11. History of regularly taking non-prescription NSAIDs (i.e. more than intermittent) within 3 months of the study
12. Known sensitivity to acetylsalicylic acid, with impaired coagulation or with ulcer, kidney or liver problems.
13. Cadiac pacemaker, metal allergy or severe needle phobia
14. Serious cardiovascular, cerebral disease, psychiatric disorder or cognitive Impairment
15. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | baseline, 2 weeks, 6 weeks, 3 months
  Change in average jaw pain intensity rated by the patient over last 24 hours and last 7 days (VAS: 0-100mm) between baseline and the following time points: 2 weeks, 6 weeks and 3 months.
  Even though patients will be treated 1-2 treatments per week for 4 weeks (up to 8 treatments total), the visual analogue score after 2 weeks of treatment, at 6 weeks (2 weeks post treatment) and at 3 months (2 months post treatment) will be compared to baseline (pre-treatment). Scores closer to 0 represent less pain.

SECONDARY OUTCOMES:
Global Rating of Perceived Change | 2 weeks, 6 weeks, 3 months
  Global rating of perceived change rated rated by the patient according to a -7 to +7 scale. More specifically, the Global Rating of Perceived Change is rated as follows:
  * A very great deal worse (-7)
  * A great deal worse (-6)
  * Quite a bit worse (-5)
  * Moderately worse (-4)
  * Somewhat worse (-3)
  * A little bit worse (-2)
  * A tiny bit worse (almost the same) (-1)
  * About the same (0)
  * A very great deal better (+7)
  * A great deal better (+6)
  * Quite a bit better (+5)
  * Moderately better (+4)
  * Somewhat better (+3)
  * A little bit better (+2)
  * A tiny bit better (almost the same) (+1)
  The patient will choose a rating (the closer to +7, the better the score / the closer to -7, the worse the score) after 2 weeks of treatment, at 6 weeks (2 weeks post-treatment) and 3 months (2 months post-treatment).
Active Pain Free Mouth Opening | baseline, 2 weeks, 6 weeks, 3 months
  Change in the distance between upper and lower central incisors after patient has opening mouth "as wide as possible" without causing pain between baseline and the following time points: 2 weeks, 6 weeks and 3 months. Measurements will be taken in mm. The greater the distance, the better the score.
  Even though patients will be treated 1-2 treatments per week for 4 weeks (up to 8 treatments total), active pain free mouth opening after 2 weeks of treatment, at 6 weeks (2 weeks post treatment) and at 3 months (2 months post treatment) will be compared to baseline (pre-treatment)
  Greater scores represent greater pain free mouth opening.

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Physiomed-lab, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided